CLINICAL TRIAL: NCT05839262
Title: Physical Exercise Guided by Active Video Games for Optimizing Clinical and Psychosocial Outcomes in Older Adults With Knee and/or Hip Osteoarthritis Under a Community-based Rehabilitation Model.
Brief Title: Active Video Games for Older Adults With Knee and/or Hip Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristian Alvarez (Other)
Collaborators: National Fund for Research and Development in Health, Chile (Other)
Responsible Party: Sponsor-Investigator, Cristian Alvarez, Associate Proffesor, Universidad Nacional Andres Bello
Organization: Universidad Nacional Andres Bello (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNAB-FCR-KINE2023B
Record Dates: First submitted 2023-03-15; First posted 2023-05-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: osteoarhrosis; elderly; exercise training; video games; public health
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial (RCT).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator: Statistical data analyst.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Conventional physical rehabilitation plus Active video games (CPR+AVG)
  Interventions: Other: Conventional physical rehabilitation plus Active video games (CPR+AVG)
- Control group (Active Comparator): Conventional physical rehabilitation alone (CPR)
  Interventions: Other: Conventional physical rehabilitation alone (CPR)

INTERVENTIONS:
Other: Conventional physical rehabilitation plus Active video games (CPR+AVG) — In each session a routine of conventional physical rehabilitation and active video games is performed. The duration is 10 weeks / 3 sessions per week (30 sessions).
  CPR+AVG: Consists of conventional exercises (aerobic, muscle strengthening, postural balance and flexibility) added to a set of interactive video games available for the Nintendo Switch console.
  Arms: Experimental group
Other: Conventional physical rehabilitation alone (CPR) — In each session a routine of conventional exercises is performed. The duration is 10 weeks / 3 sessions per week (30 sessions).
  CPR: Conventional exercises (aerobic, muscle strengthening, postural balance and flexibility).
  Arms: Control group

SUMMARY:
Population aging is currently an issue of primary relevance, constituting an enormous challenge for institutions and society. On the other hand, osteoarthritis (OA) is the most prevalent arthropathy in the elderly, strongly related to loss of functional capacity, limitation of daily activities, increased musculoskeletal pain, and deterioration of quality of life. More specifically, knee and hip OA represent a significant burden for health systems, and in Chile, they are among the ten most frequent diseases in the elderly. The technological development of the last decades has allowed the incorporation of several therapeutic alternatives for the intervention of the elderly, such as virtual reality, which allows interaction with multiple digital environments. Active video games (AVG) or exergames, carried out through commercial non-immersive virtual reality systems, have been proposed as a feasible, innovative, and entertaining alternative to optimize conventional physical rehabilitation (CPR). AVG in healthy older people and those with neurocognitive conditions effectively improves clinical and psychosocial outcomes. However, it has been recommended to advance the study of the effects of AVGs in people with musculoskeletal pathologies, such as knee and hip OA. Accordingly, the purpose is to analyze the effects of an AVG-guided physical exercise protocol adjunct to CPR on functional mobility in older adults with knee and/or hip OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is highly prevalent, and its incidence increases with aging populations. OA is characterized by articular cartilage degeneration, stiffness, inflammation, and musculoskeletal pain. In addition, the associated deterioration of health-related quality of life may influence therapeutic adherence and progression to future joint replacement. It appears that symptoms rather than structural impairment determine the risk of falling in older people with OA, so pain, loss of strength, and postural balance are underlying mechanisms for both falls and the clinical picture of OA itself. Moreover, the psychosocial sequelae are often underestimated because OA and pain are usually considered benign and unavoidable consequences of aging.

Physical exercise in people with knee and hip OA improves clinical aspects and psychosocial aspects such as self-efficacy, social function, and reduction of depression and isolation, among others. Adherence to exercise is fundamental and is closely related to user satisfaction. There are several barriers to physical exercise by older adults, such as lack of social support, transportation problems, and prioritization of basic needs; however, a determining factor is lack of motivation. In this regard, a study indicates that in Latin America, lack of motivation is among the main reasons for abandoning physical exercise.

The technological development of the last decades has allowed the incorporation of virtual reality into the healthcare field, favoring user motivation. Virtual reality is an experience based on the interactive digital simulation of environments and objects. These systems are categorized as non-immersive, semi-immersive, and immersive. Non-immersive systems use monitors or television screens, semi-immersive systems use panoramic screens to enhance the immersive experience, and immersive systems use head-mounted displays or multi-projected environments that generate a strong sense of immersion. It has been posited that the cost and expertise required to operate immersive systems may hinder their widespread use in clinical settings. In addition, the immersive sensation could produce symptoms such as visual fatigue and dizziness (cybersickness). On the other hand, non-immersive systems using commercially available home consoles are now considered an attractive and more accessible alternative to more sophisticated immersive systems.

Unlike traditional video games that use a standard command or joystick, active video games (AVGs) (also called exergames) use motion monitoring systems such as accelerometers, gyroscopes, haptic technology, and video capture. AVGs have been defined as a "combination of video game technologies and exercise routines to motivate physical activity among individuals or groups," recognizing that exercise in older people requires a greater understanding of the complexity of interaction with computer systems.

Conventional physical rehabilitation (CPR) consists of traditional physical exercises that improve functional capacity. Over the past few years, it has been suggested that incorporating AVGs into CPR can optimize clinical and psychosocial outcomes in the elderly. AVGs have been reported to promote improvements in functional mobility, coordination, muscle strength, and cognitive function in older people. In addition, AVGs improve walking ability and postural balance, as well as social well-being (perception of loneliness, social connectedness, and positive attitudes). However, this research has focused on healthy elderly and patients with neurocognitive pathologies. On the other hand, little information is available on older people with musculoskeletal conditions such as OA. In this regard, a systematic review conducted in patients with knee and/or hip OA indicates that the evidence is insufficient and inconclusive regarding the effectiveness of AVGs. Moreover, one study concludes that AVGs are a feasible and acceptable intervention for patients with knee OA. Interestingly, both studies raise the benefits and potential of AVGs in this population, urging further clinical trials.

Research question: In older adults with knee and/or hip OA. Is AVG-guided physical exercise adjunct to CPR more effective than CPR alone in improving clinical and psychosocial outcomes?

Working hypothesis: In older adults with knee and/or hip OA, AVG-guided physical exercise adjunct to CPR is more effective than CPR alone in improving clinical and psychosocial outcomes.

General objective: To determine the effects of an AVG-guided physical exercise program adjunct to CPR on clinical and psychosocial outcomes in older adults with knee and/or hip OA attended at a community-based family health center.

Specific objectives:

1. To characterize the study sample from sociodemographic, anthropometric, clinical, and psychosocial perspectives.
2. To compare the results of the primary outcome (functional mobility) and secondary outcomes between the study groups (experimental and control) in the different instances of outcome measurement.
3. To evaluate the clinical significance of the interventions and the clinical relevance of the interventions as perceived by the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 and ≤84 years.
* Diagnosis of mild or moderate OA of the knee and/or hip.
* Independent walking capacity of at least 15 meters.

Exclusion Criteria:

* Inability to interact with active video games.
* Undergoing treatment with opioids or other medications with a potential influence on the outcomes of interest.
* <13 points in the abbreviated version of the Mini-Mental State Examination (MMSE-EFAM).
* OA associated with infectious, autoimmune, fractures or surgery.
* Participate or have participated in another physical-cognitive rehabilitation program during the last 3 months.

Ages: 60 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Functional mobility. | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  Timed Up and Go (TUG). Number of seconds required to get up from seated position, walk 3 m, turn, and return to seated position on chair.

SECONDARY OUTCOMES:
Change in Lower body strength. | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  30-s chair stand. Number of full stands in 30 s with arms folded across chest
Change in Upper body strength. | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  30-s arm curl. Number of bicep curls in 30 s holding hand weight (women 5 lb; men 8 lb)
Change in Aerobic endurance. | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  2-min step test. Number of full steps completed in 2 min,raising each knee to point midway between patella and iliac crest (score is number of times right knee reaches target)
Change in Lower body flexibility | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  Chair sit-and-reach. From sitting position at front of chair, with leg extended and hands reaching toward toes, number of inches (+or - ) from extended fingers to tip of toe
Change in Upper body flexibility. | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  Back scratch. With one hand reaching over shoulder and one up middle of back, number of inches between extended middle fingers (+ or - )
Change in Hand grip strength | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  Number of kg measured with a Jamar dynamometer.
Change in Functional disability. | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  Western Ontario McMaster Osteoarthritis Index (WOMAC) questionnaire. Score obtained on the scale of items grouped into 3 dimensions: pain, stiffness and difficulty in performing tasks. Scores range from 0 to 96, where 0 represents the best health status and 96 the worst possible status.
Change in Cognitive performance. | Three-time points. Baseline (pre-intervention); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  Montreal Cognitive Assessment (MoCA) test. Score obtained in the development of the tests. It considers executive functions, attention, abstraction, memory, language, viso-constructive abilities, calculation and orientation. MoCA scores range from 0 to 30; higher scores indicate a better cognitive performance.
Change in Pain intensity. | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  Visual Analog Scale (VAS). 100 mm straight line with two labels ("no pain" and "worst possible pain") at each end.
Change in Pressure pain threshold | Five-time points. Baseline (pre-intervention); at week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  Wagner® FPX-25 algometer. It is expressed in kilogram/cm2.
Change in Health-related quality of life | Three-time points. Baseline (pre-intervention); and week 10 (after 30 sessions from baseline). In addition, four weeks after the completion of the intervention.
  SF-12v2 Chile-Spanish Questionnaire. Score from 0-100 points. Assessment of 8 dimensions (physical functioning [PF], role-physical [RP], bodily pain [BP], general health [GH], vitality [VT], social functioning [SF], role-emotional [RE], and mental health [MH]), and two summary scores (physical component summary [PCS] and mental component summary [MCS]).
Adherence to treatment | One-time point. At week 10 (after 30 sessions from baseline).
  Number of effective assistances at the end of treatment. A participant with an attendance ≥2/3 of the total (30 sessions) is considered "adherent" (≥20 sessions).
Change in User satisfaction | Three-time points. At week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline).
  The average score of 3 questions (overall level of satisfaction, expectation fulfillment, and recommendations to others) using a scale of 1 to 7 points, where 1 is the worst evaluation, and 7 is the best evaluation.
Change in Therapeutic alliance | Three-time points. At week 4 (after ten sessions from baseline); at week 7 (after 20 sessions from baseline); and week 10 (after 30 sessions from baseline).
  Subscale of the Pain Rehabilitation Expectations Scale (PRES). The score ranges from 1 to 44; a higher score is a higher therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Cristhian Mendoza S., PhD, Study Chair — Universidad San Sebastian; Claudio Carvajal P., PhD, Study Director — Universidad San Sebastian; Jorge Fuentes C., PhD, Study Director — Universidad Católica del Maule; Camila Riquelme B., Study Director — Universidad Andrés Bello
Locations (1):
- Centro de Salud Familiar (CESFAM) Lorenzo Arenas, Concepción, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spitaels D, Mamouris P, Vaes B, Smeets M, Luyten F, Hermens R, Vankrunkelsven P. Epidemiology of knee osteoarthritis in general practice: a registry-based study. BMJ Open. 2020 Jan 20;10(1):e031734. doi: 10.1136/bmjopen-2019-031734. PMID 31964664
- [Background] Rosen J, Niazi F, Dysart S. Cost-Effectiveness of Treating Early to Moderate Stage Knee Osteoarthritis with Intra-articular Hyaluronic Acid Compared to Conservative Interventions. Adv Ther. 2020 Jan;37(1):344-352. doi: 10.1007/s12325-019-01142-x. Epub 2019 Nov 18. PMID 31735982
- [Background] Ho KW, Pong G, Poon WC, Chung KY, Kwok YY, Chiu KH. Progression of health-related quality of life of patients waiting for total knee arthroplasty. J Eval Clin Pract. 2021 Feb;27(1):69-74. doi: 10.1111/jep.13388. Epub 2020 Mar 22. PMID 32202045
- [Background] Mat S, Ng CT, Tan MP. Influence of hip and knee osteoarthritis on dynamic postural control parameters among older fallers. J Rehabil Med. 2017 Mar 6;49(3):258-263. doi: 10.2340/16501977-2202. PMID 28218341
- [Background] Manlapaz DG, Sole G, Jayakaran P, Chapple CM. Risk Factors for Falls in Adults with Knee Osteoarthritis: A Systematic Review. PM R. 2019 Jul;11(7):745-757. doi: 10.1002/pmrj.12066. Epub 2019 Mar 28. PMID 30609282
- [Background] Hurley M, Dickson K, Hallett R, Grant R, Hauari H, Walsh N, Stansfield C, Oliver S. Exercise interventions and patient beliefs for people with hip, knee or hip and knee osteoarthritis: a mixed methods review. Cochrane Database Syst Rev. 2018 Apr 17;4(4):CD010842. doi: 10.1002/14651858.CD010842.pub2. PMID 29664187
- [Background] Klaps S, Haesevoets S, Verbunt J, Koke A, Janssens L, Timmermans A, Verbrugghe J. The Influence of Exercise Intensity on Psychosocial Outcomes in Musculoskeletal Disorders: A Systematic Review. Sports Health. 2022 Nov-Dec;14(6):859-874. doi: 10.1177/19417381221075354. Epub 2022 Mar 4. PMID 35243924
- [Background] Hawley-Hague H, Horne M, Skelton DA, Todd C. Review of how we should define (and measure) adherence in studies examining older adults' participation in exercise classes. BMJ Open. 2016 Jun 23;6(6):e011560. doi: 10.1136/bmjopen-2016-011560. PMID 27338884
- [Background] Room J, Hannink E, Dawes H, Barker K. What interventions are used to improve exercise adherence in older people and what behavioural techniques are they based on? A systematic review. BMJ Open. 2017 Dec 14;7(12):e019221. doi: 10.1136/bmjopen-2017-019221. PMID 29247111
- [Background] Franco MR, Tong A, Howard K, Sherrington C, Ferreira PH, Pinto RZ, Ferreira ML. Older people's perspectives on participation in physical activity: a systematic review and thematic synthesis of qualitative literature. Br J Sports Med. 2015 Oct;49(19):1268-76. doi: 10.1136/bjsports-2014-094015. Epub 2015 Jan 13. PMID 25586911
- [Background] Cigarroa I, Zapata-Lamana R, Leiva-Gajardo G, Vasquez E, Parrado-Romero E, Vásquez-Gomez J, et al. Adherence characteristics and reasons for abandonment of physical exercise-based interventions in older adults in Latin America: A scoping review (Características de la adherencia y motivos del abandono de las intervenciones basadas en el ejercicio físic. Retos. 2022 Apr 1;44:10-26.
- [Background] Torner J, Skouras S, Molinuevo JL, Gispert JD, Alpiste F. Multipurpose Virtual Reality Environment for Biomedical and Health Applications. IEEE Trans Neural Syst Rehabil Eng. 2019 Aug;27(8):1511-1520. doi: 10.1109/TNSRE.2019.2926786. Epub 2019 Jul 4. PMID 31283482
- [Background] Mirelman A, Maidan I, Shiratzky SS, Hausdorff JM. Virtual Reality Training as an Intervention to Reduce Falls. In: Montero-Odasso M, Camicioli R, editors. Falls and Cognition in Older Persons: Fundamentals, Assessment and Therapeutic Options. Cham: Springer International Publishing; 2020. p. 309-21.
- [Background] Marston HR, Smith ST. Interactive Videogame Technologies to Support Independence in the Elderly: A Narrative Review. Games Health J. 2012 Apr;1(2):139-52. doi: 10.1089/g4h.2011.0008. PMID 26193189
- [Background] Zheng L, Li G, Wang X, Yin H, Jia Y, Leng M, Li H, Chen L. Effect of exergames on physical outcomes in frail elderly: a systematic review. Aging Clin Exp Res. 2020 Nov;32(11):2187-2200. doi: 10.1007/s40520-019-01344-x. Epub 2019 Sep 13. PMID 31520334
- [Background] Kappen DL, Mirza-Babaei P, Nacke LE. Older Adults' Physical Activity and Exergames: A Systematic Review. International Journal of Human-Computer Interaction. 2019 Jan 20;35(2):140-67.
- [Background] Levine M, McElroy K, Stakich V, Cicco J. Comparing conventional physical therapy rehabilitation with neuromuscular electrical stimulation after TKA. Orthopedics. 2013 Mar;36(3):e319-24. doi: 10.3928/01477447-20130222-20. PMID 23464951
- [Background] Tousignant M, Corriveau H, Roy PM, Desrosiers J, Dubuc N, Hebert R. Efficacy of supervised Tai Chi exercises versus conventional physical therapy exercises in fall prevention for frail older adults: a randomized controlled trial. Disabil Rehabil. 2013 Aug;35(17):1429-35. doi: 10.3109/09638288.2012.737084. Epub 2012 Nov 20. PMID 23167499
- [Background] Li J, Erdt M, Chen L, Cao Y, Lee SQ, Theng YL. The Social Effects of Exergames on Older Adults: Systematic Review and Metric Analysis. J Med Internet Res. 2018 Jun 28;20(6):e10486. doi: 10.2196/10486. PMID 29954727
- [Background] Collado-Mateo D, Merellano-Navarro E, Olivares PR, Garcia-Rubio J, Gusi N. Effect of exergames on musculoskeletal pain: A systematic review and meta-analysis. Scand J Med Sci Sports. 2018 Mar;28(3):760-771. doi: 10.1111/sms.12899. Epub 2017 May 22. PMID 28452070
- [Background] Cacciata M, Stromberg A, Lee JA, Sorkin D, Lombardo D, Clancy S, Nyamathi A, Evangelista LS. Effect of exergaming on health-related quality of life in older adults: A systematic review. Int J Nurs Stud. 2019 May;93:30-40. doi: 10.1016/j.ijnurstu.2019.01.010. Epub 2019 Feb 10. PMID 30861452
- [Background] Viana RB, de Oliveira VN, Dankel SJ, Loenneke JP, Abe T, da Silva WF, Morais NS, Vancini RL, Andrade MS, de Lira CAB. The effects of exergames on muscle strength: A systematic review and meta-analysis. Scand J Med Sci Sports. 2021 Aug;31(8):1592-1611. doi: 10.1111/sms.13964. Epub 2021 Apr 15. PMID 33797115
- [Background] Bevilacqua R, Maranesi E, Riccardi GR, Donna VD, Pelliccioni P, Luzi R, Lattanzio F, Pelliccioni G. Non-Immersive Virtual Reality for Rehabilitation of the Older People: A Systematic Review into Efficacy and Effectiveness. J Clin Med. 2019 Nov 5;8(11):1882. doi: 10.3390/jcm8111882. PMID 31694337
- [Background] Reis E, Postolache G, Teixeira L, Arriaga P, Lima ML, Postolache O. Exergames for motor rehabilitation in older adults: an umbrella review. Physical Therapy Reviews. 2019 Jul 4;24(3-4):84-99.
- [Background] Corregidor-Sanchez AI, Segura-Fragoso A, Rodriguez-Hernandez M, Criado-Alvarez JJ, Gonzalez-Gonzalez J, Polonio-Lopez B. Can exergames contribute to improving walking capacity in older adults? A systematic review and meta-analysis. Maturitas. 2020 Feb;132:40-48. doi: 10.1016/j.maturitas.2019.12.006. Epub 2019 Dec 9. PMID 31883662
- [Background] Fang Q, Ghanouni P, Anderson SE, Touchett H, Shirley R, Fang F, Fang C. Effects of Exergaming on Balance of Healthy Older Adults: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Games Health J. 2020 Feb;9(1):11-23. doi: 10.1089/g4h.2019.0016. Epub 2019 Dec 3. PMID 31800322
- [Background] Ismail NA, Hashim HA, Ahmad Yusof H. Physical Activity and Exergames Among Older Adults: A Scoping Review. Games Health J. 2022 Feb;11(1):1-17. doi: 10.1089/g4h.2021.0104. Epub 2021 Dec 1. PMID 34851732
- [Background] Janhunen M, Karner V, Katajapuu N, Niiranen O, Immonen J, Karvanen J, Heinonen A, Aartolahti E. Effectiveness of Exergame Intervention on Walking in Older Adults: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Phys Ther. 2021 Sep 1;101(9):pzab152. doi: 10.1093/ptj/pzab152. PMID 34160022
- [Background] Swinnen N, Vandenbulcke M, Vancampfort D. Exergames in people with major neurocognitive disorder: a systematic review. Disabil Rehabil Assist Technol. 2022 May;17(4):376-389. doi: 10.1080/17483107.2020.1785566. Epub 2020 Jul 22. PMID 32697614
- [Background] Prosperini L, Tomassini V, Castelli L, Tacchino A, Brichetto G, Cattaneo D, Solaro CM. Exergames for balance dysfunction in neurological disability: a meta-analysis with meta-regression. J Neurol. 2021 Sep;268(9):3223-3237. doi: 10.1007/s00415-020-09918-w. Epub 2020 May 23. PMID 32447551
- [Background] Wang B, Shen M, Wang YX, He ZW, Chi SQ, Yang ZH. Effect of virtual reality on balance and gait ability in patients with Parkinson's disease: a systematic review and meta-analysis. Clin Rehabil. 2019 Jul;33(7):1130-1138. doi: 10.1177/0269215519843174. Epub 2019 Apr 24. PMID 31016994
- [Background] Zhao Y, Feng H, Wu X, Du Y, Yang X, Hu M, Ning H, Liao L, Chen H, Zhao Y. Effectiveness of Exergaming in Improving Cognitive and Physical Function in People With Mild Cognitive Impairment or Dementia: Systematic Review. JMIR Serious Games. 2020 Jun 30;8(2):e16841. doi: 10.2196/16841. PMID 32602841
- [Background] Byra J, Czernicki K. The Effectiveness of Virtual Reality Rehabilitation in Patients with Knee and Hip Osteoarthritis. J Clin Med. 2020 Aug 14;9(8):2639. doi: 10.3390/jcm9082639. PMID 32823832
- [Background] Manlapaz DG, Sole G, Jayakaran P, Chapple CM. Exergaming to improve balance and decrease the risk of falling in adults with knee osteoarthritis: a mixed-methods feasibility study. Physiother Theory Pract. 2022 Nov;38(13):2428-2440. doi: 10.1080/09593985.2021.1952670. Epub 2021 Jul 19. PMID 34280069
- [Background] Lin HT, Li YI, Hu WP, Huang CC, Du YC. A Scoping Review of The Efficacy of Virtual Reality and Exergaming on Patients of Musculoskeletal System Disorder. J Clin Med. 2019 Jun 4;8(6):791. doi: 10.3390/jcm8060791. PMID 31167435
- [Derived] Guede-Rojas F, Mendoza C, Rodriguez-Lagos L, Soto-Martinez A, Ulloa-Diaz D, Jorquera-Aguilera C, Carvajal-Parodi C. Effects of Non-Immersive Virtual Reality Exercise on Self-Reported Pain and Mechanical Hyperalgesia in Older Adults with Knee and Hip Osteoarthritis: A Secondary Analysis of a Randomized Controlled Trial. Medicina (Kaunas). 2025 Jun 21;61(7):1122. doi: 10.3390/medicina61071122. PMID 40731752

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT05839262/Prot_SAP_000.pdf